CLINICAL TRIAL: NCT04267380
Title: Compare Effectiveness of Tofacitinib 11 mg QD to Tofacitinib 5 mg BID
Brief Title: A Study To Compare The Effectiveness Of Tofacitinib 11 Mg Once A Day To Tofacitinib 5 Mg Twice A Day
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921359
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Arthritis Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corrona US RA Registry 11 mg: patients with RA who have been exposed to tofacitinib 11 mg QD tablet
- Corrona US RA Registry 5 mg: patients with RA who have been exposed to tofacitinib 5 mg BID tablet

SUMMARY:
It is hypothesized that patients prescribed tofacitinib 11 mg Modified Release (MR) formulation once daily (QD) will achieve similar benefit to those prescribed tofacitinib 5 mg twice a day (BID) dosage in real world use. This study will therefore seek to compare the effectiveness of the MR 11 mg QD regimen to the IR 5 mg BID regimen for the treatment of RA in a real-world registry of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* All US Corrona RA Registry patients who initiated tofacitinib 5 mg twice a day (BID) or tofacitinib 11 mg once daily (QD) after it became available in February 2016
* Patients must have a follow-up visit at 6 months (+/- 3 months) after tofacitinib initiation. These 6 month visits are part of routine practice and is not associated with this protocol.
* Patients must have a valid clinical disease activity index (CDAI) at initiation and at 6-month follow-up visit

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients prescribed Tofacitinib in routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cohen SB, Greenberg JD, Harnett J, Madsen A, Smith TW, Gruben D, Zhang R, Lukic T, Woolcott J, Dandreo KJ, Litman HJ, Blachley T, Lenihan A, Chen C, Rivas JL, Dougados M. Real-World Evidence to Contextualize Clinical Trial Results and Inform Regulatory Decisions: Tofacitinib Modified-Release Once-Daily vs Immediate-Release Twice-Daily for Rheumatoid Arthritis. Adv Ther. 2021 Jan;38(1):226-248. doi: 10.1007/s12325-020-01501-z. Epub 2020 Oct 9. PMID 33034006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was retrospective study of participants with rheumatoid arthritis (RA) who were tofacitinib initiators (first ever use of tofacitinib as reported by rheumatologist) on or after February 2016. Such participants were identified and their data was retrieved from United States (US) Corrona RA Registry database and assessed in this study.
Groups:
- Tofacitinib Modified Release (MR) 11mg QD: Participants with RA who initiated Tofacitinib 11 milligram (mg) MR tablet, orally, once daily (QD), after February 2016 and followed up for 6 months after tofacitinib initiation were included in this study. Their information as per US Corrona RA Registry database for approximately 3.7 years from February 2016 to end of September 2019 was assessed in this study. Baseline in the study is defined as the time of tofacitinib initiation.
- Tofacitinib Immediate Release (IR) 5 mg BID: Participants with RA who initiated Tofacitinib 5 mg IR tablet, orally, twice daily (BID), on or after February 2016 and followed up for 6 months after tofacitinib initiation were included in this study. Their information as per US Corrona RA Registry database for approximately 3.7 years from February 2016 to end of September 2019 was assessed in this study. Baseline in the study is defined as the time of tofacitinib initiation.
Period: Overall Study
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Started | 149 | 149
Completed | 149 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants included in the study.
Groups:
- Tofacitinib Modified Release (MR) 11mg QD: Participants with RA who initiated Tofacitinib 11mg MR tablet, orally, QD, after February 2016 and followed up for 6 months after tofacitinib initiation were included in this study. Their information as per US Corrona RA Registry database for approximately 3.7 years from February 2016 to end of September 2019 was assessed in this study. Baseline in the study is defined as the time of tofacitinib initiation.
- Tofacitinib Immediate Release (IR) 5 mg BID: Participants with RA who initiated Tofacitinib 5 mg IR tablet, orally, BID, on or after February 2016 and followed up for 6 months after tofacitinib initiation were included in this study. Their information as per US Corrona RA Registry database for approximately 3.7 years from February 2016 to end of September 2019 was assessed in this study. Baseline in the study is defined as the time of tofacitinib initiation.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID | Total
Number analyzed (Participants) | 149 | 149 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (12.0) | 60.8 (11.5) | 60.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 117 | 237
  Male | 29 | 32 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 129 | 130 | 259
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Minimally Clinically Important Difference (MCID) Improvement From Baseline Upto 6 Months
Description: MCID improvement assessed based on Clinical disease activity index (CDAI). CDAI: numerical sum of 4 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient global assessment (PtGA) and physician global assessment (PGA) assessed on 0-10 centimeter (cm) Visual analogue scale (VAS); CDAI total score = 0-76, higher scores=greater affection due to disease activity (DA). CDAI less than or equal to (<=) 2.8 indicates disease remission, greater than (>) 2.8 to 10 = low DA, >10 to 22 = moderate DA, and >22 = high DA. MCID improvement defined by difference in CDAI from baseline (at time of tofacitinib initiation) to 6 month visit. Participants were considered to show improvement from baseline on 3 cut points (1) greater than or equal (>=) to 2 (for participants in low DA at baseline); (2) >= 6 (moderate DA at baseline, and (3) >= 11 (high DA at baseline). Here, overall number of participants who showed improvement have been reported.
Time Frame: Baseline Up to 6 Months
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 38 | 33
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.73, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Month 6
Description: CDAI is the numerical sum of 4 outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 to 10 cm VAS; CDAI total score = 0 to 76, higher scores=greater affection due to disease activity. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Here, all participants who achieved remission (CDAI <=2.8) at Month 6 have been reported.
Time Frame: Baseline, Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
units on a scale
  Baseline | 16.4 (12.2) | 17.9 (14.6)
  Change at Month 6 | -2.19 (13.08) | -2.12 (12.74)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.97, t-test, 2 sided

3. Secondary Outcome: Number of Participants Achieving Remission at Month 6 (All Participants)
Description: as for outcome 2
Time Frame: Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 13 | 8
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.26, Chi-squared

4. Secondary Outcome: Number of Participants Achieving Remission at Month 6 (For Participants With Baseline CDAI >2.8)
Description: CDAI is the numerical sum of 4 outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 to 10 cm VAS; CDAI total score = 0 to 76, higher scores=greater affection due to disease activity. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Here, only those participants who had baseline CDAI greater than 2.8, and who achieved remission (CDAI <= 2.8) at Month 6 have been reported.
Time Frame: Month 6
Population: Analysis was performed on only those participants who had baseline CDAI greater than 2.8. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 139 | 140
Participants | 8 | 4
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.23, Chi-squared

5. Secondary Outcome: Number of Participants Achieving Low Disease Activity at Month 6 (All Participants)
Description: CDAI is the numerical sum of 4 outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 to 10 cm VAS; CDAI total score = 0 to 76, higher scores=greater affection due to disease activity. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Here, all participants who achieved low disease activity (CDAI > 2.8 to 10) at Month 6 have been reported.
Time Frame: Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 54 | 46
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.33, Chi-squared

6. Secondary Outcome: Number of Participants Achieving Low Disease Activity at Month 6 (Participants With Baseline CDAI >10)
Description: CDAI is the numerical sum of 4 outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 to 10 cm VAS; CDAI total score = 0 to 76, higher scores=greater affection due to disease activity. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Here, only those participants who had baseline CDAI greater than 10, and who achieved low disease activity (CDAI > 2.8 to 10) at Month 6 have been reported.
Time Frame: Month 6
Population: Analysis was performed on only those participants who had baseline CDAI greater than 10. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 96 | 94
Participants | 28 | 17
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.07, Chi-squared

7. Secondary Outcome: Number of Participants With Decrease From Baseline in Modified Health Assessment Questionnaire (mHAQ) Score at Month 6
Description: Modified HAQ: participant-reported questionnaire for the assessment of ability to perform tasks due to rheumatoid arthritis. It comprised of 8 questions on 8 categories of daily living activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and common activities over past week before specified time point. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Participants who had a baseline mHAQ score of >=0.25 were evaluable for this outcome measure and number of participants who had decrease from baseline in mHAQ score at Month 6 were reported.
Time Frame: Month 6
Population: Analysis was performed on participants who had a baseline mHAQ score of >=0.25. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 99 | 97
Participants | 24 | 26
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.68, Chi-squared

8. Secondary Outcome: Number of Participants With Decrease From Baseline in Health Assessment Questionnaire (HAQ) Score at Month 6
Description: HAQ: participant-reported questionnaire for the assessment of rheumatoid arthritis. It comprised of 20 questions in 8 categories of activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and activities over past week. Each activity was assessed on a 4-point Likert scale from 0 to 3, where 0 = without difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Participants who had a baseline HAQ score of >=0.22 were evaluable for this outcome measure and number of participants who had decrease from baseline in HAQ score at Month 6 were reported.
Time Frame: Month 6
Population: Analysis was performed on participants who had a baseline HAQ score of >=0.22. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 122 | 124
Participants | 24 | 27
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.68, Chi-squared

9. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Month 6: Dichotomous Variable
Time Frame: Baseline, Month 6
Population: Data for change from baseline in HAQ score as 'dichotomous variable' was not collected, as this outcome measure was inappropriately included in protocol specified secondary outcomes.
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Modified Health Assessment Questionnaire (mHAQ) Score at Month 6
Description: Modified HAQ: participant-reported questionnaire for the assessment of ability to perform tasks due to rheumatoid arthritis. It comprised of 8 questions in 8 categories of daily living activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and common activities over past week. Eight item were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for mHAQ. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 139 | 144
units on a scale | -0.02 (0.41) | -0.06 (0.38)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.45, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ) Score at Month 6
Description: HAQ: participant-reported questionnaire for the assessment of rheumatoid arthritis. It comprised of 20 questions in 8 categories of activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and activities over past week. Each activity was assessed on a 4-point Likert scale from 0 to 3, where 0 = without difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for HAQ. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 130 | 133
units on a scale | -0.03 (0.50) | -0.07 (0.46)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.53, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Modified Disease Activity Score Based on 28-joints Count (mDAS28) at Month 6
Description: Modified DAS28: Indicator of disease activity calculated as weighted average of six components: tender joint counts (TJC), swollen joint counts (SJC), mHAQ measure of disease activity, participant reported pain, physician reported global health assessment (PGA) and participant reported global health assessment (PtGA). TJC and SJC calculated using 28 joints count; mHAQ scored on a scale of 0 to 3 (0 = least difficulty, 3 = extreme difficulty); participant reported pain scored on a scale of 0 to 100 (0 = no pain, 100= pain as bad as it could be); PGA and PtGA recorded on a visual analog scale (VAS) of 0 millimeter (mm) to 100 mm (0 = no disease activity and 100=high disease activity). Transformed mDAS28 score ranged from 0 to 9.4, where higher scores indicated more disease activity.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for mDAS28. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 139 | 144
units on a scale
  Baseline | 4.1 (1.4) | 4.2 (1.5)
  Change at Month 6 | -0.23 (1.41) | -0.20 (1.34)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.86, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count (DAS28) Erythrocyte Sedimentation Rate (ESR) at Month 6
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (millimeters per hour) and PtGA recorded on 100mm VAS (scores ranging 0 [very well] to 100 mm [extremely bad]). DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln(ESR [mm/hour] + 0.014*PtGA [mm]; where, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for DAS28 (ESR). Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 68 | 71
units on a scale
  Baseline | 3.9 (1.6) | 4.0 (1.6)
  Change at Month 6 | -0.17 (1.80) | -0.10 (1.70)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.83, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count (DAS28) C- Reactive Protein (CRP) at 6 Month
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis. DAS28 (CRP) was calculated from SJC and TJC using 28 joints count, CRP (milligrams per liter [mg/L]) and PtGA on a 100 mm VAS (VAS: scores ranging from 0 mm [very well] to 100 mm [worst], higher scores indicate worse health condition). DAS28 (CRP) was calculated as = 0.56*sqrt(TJC28) + 0.28*sqrt(SJC28) + 0.36*ln(CRP in mg/L +1) + 0.014*PtGA in mm+ 0.96.Total DAS28 (CRP) score range: 0 (none) to 9.4 (extreme disease activity), higher score indicated more disease activity.
Time Frame: Baseline, 6 months
Population: Analysis was performed on participants included in the study who were evaluable for DAS28 (CRP). Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 80 | 72
units on a scale
  Baseline | 3.6 (1.4) | 3.9 (1.5)
  Change at Month 6 | -0.22 (1.57) | -0.33 (1.56)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.67, t-test, 2 sided

15. Secondary Outcome: Change From Baseline in Participant Pain Score at Month 6
Description: Participants were asked the following question to answer on a numeric rating scale (NRS): "How much pain have you had because of your arthritis in the past week?" The scale ranged from 0-100, where 0=no pain and 100=pain as bad as it could be. Higher scores indicated worsening of condition.
Time Frame: Baseline, Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
units on a scale
  Baseline | 48.2 (28.6) | 48.3 (27.4)
  Change at Month 6 | -1.30 (28.56) | -0.78 (21.73)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.86, t-test, 2 sided

16. Secondary Outcome: Change From Baseline in Participant Fatigue Score at Month 6
Description: Participants were asked the following question to answer on NRS: "How much of a problem has unusual fatigue of tiredness been for you in the past week?" The scale ranged from 0-100, where 0=no fatigue and 100=fatigue as bad as it could be. Higher scores indicated worsening of condition.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for fatigue score. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 146 | 148
units on a scale
  Baseline | 48.6 (30.1) | 50.6 (29.9)
  Change at Month 6 | -0.04 (28.08) | -0.86 (22.29)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.78, t-test, 2 sided

17. Secondary Outcome: Change From Baseline in European Quality of Life- 5 Dimension (EQ-5D) Index at Month 6
Description: EQ-5D index: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. It assesses level of current health in 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension had 3 levels: no problems (1), some problems (2) and severe problems (3). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range 0 to 1, where 0=death and 1=perfect health; higher score indicates a better health state.
Time Frame: Baseline, Month 6
Population: Analysis was performed on participants included in the study who were evaluable for EQ-5D score. Hence, "Overall Number of Participants Analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 126 | 122
units on a scale
  Baseline | 0.7 (0.2) | 0.7 (0.2)
  Change at Month 6 | 0.00 (0.17) | 0.00 (0.19)
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.99, t-test, 2 sided

18. Secondary Outcome: Number of Participants Achieving Modified American College of Rheumatology 20% (mACR20) Response
Description: mACR20 response: >= 20 percent (%) improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain) ; 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 14 | 23
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.11, Chi-squared

19. Secondary Outcome: Number of Participants Achieving Modified American College of Rheumatology 50% (mACR50) Response
Description: mACR50 response: >= 50% improvement in tender and swollen joint count and 50% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain) ; 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 8 | 10
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.63, Chi-squared

20. Secondary Outcome: Number of Participants Achieving Modified American College of Rheumatology 70% (mACR70) Response
Description: mACR70 response: >= 70% improvement in tender and swollen joint count and 70% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain) ; 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function).
Time Frame: Month 6
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
Number analyzed (Participants) | 149 | 149
Participants | 5 | 2
Statistical Analysis 1: Comparison: Tofacitinib Modified Release (MR) 11mg QD vs Tofacitinib Immediate Release (IR) 5 mg BID; Test type: Superiority; p = 0.25, Chi-squared

ADVERSE EVENTS:
Time Frame: Not collected
Description: Due to non-interventional nature of study, safety data was not planned to be collected during the study.
Arm/Group | Tofacitinib Modified Release (MR) 11mg QD | Tofacitinib Immediate Release (IR) 5 mg BID
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04267380/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04267380/SAP_001.pdf